CLINICAL TRIAL: NCT03246828
Title: Investigating Glucagon Secretion in HNF1-alpha and HNF4-alpha MODY
Brief Title: Glucagon in MODY (Maturity Onset Diabetes of the Young)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12538
Record Dates: First submitted 2017-07-04; First posted 2017-08-11 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: MODY1; MODY3
Keywords: gliclazide; glucagon; diabetes
MeSH Terms: conditions — Maturity-Onset Diabetes of the Young, Type 1; Maturity-Onset Diabetes of the Young, Type 3; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Omission of gliclazide (Experimental)
  Interventions: Other: Omission of gliclazide

INTERVENTIONS:
Other: Omission of gliclazide — Participants will stop taking gliclazide for 3 days. Data from the OGTT will be compared with that prior to stopping the medication.

SUMMARY:
The aim of this study is to determine whether fasting and post-prandial glucagon secretion is suppressed by gliclazide in patients with HNF1-/4-alpha MODY. Participants will undergo an oral glucose tolerance test (OGTT) before and after omitting their gliclazide medication for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HNF1-alpha or HNF4-alpha MODY.
* Currently on gliclazide treatment

Exclusion Criteria:

* Currently taking any anti-diabetic medication other than gliclazide and metformin
* Oral steroid treatment 30 days prior to the start or at any time during the study period.
* Known malignancy or any other condition or circumstance which, in the opinion of the investigator, would affect the patient's ability to participate in the protocol.
* Felt to be unsuitable to participate in the study in the opinion of the Chief Investigator.
* Currently participating in a clinical trial involving an anti-diabetic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Change in plasma glucagon from baseline (0min) | 0min, 30min, 60min, 90min and 120min during 75g oral glucose tolerance test.
  Change in the concentration of plasma glucagon from baseline during an oral glucose tolerance test (OGTT), while on gliclazide and after a washout period.

SECONDARY OUTCOMES:
Change in plasma c-peptide from baseline (0min) | 0min, 30min, 60min, 90min and 120min during 75g oral glucose tolerance test.
  To determine whether changes in post-prandial glucagon levels correlate with changes in c-peptide levels in HNF1-/4-alpha MODY patients on and off gliclazide.
Change in plasma non-esterified fatty acids (NEFA) from baseline (0min) | 0min, 30min, 60min, 90min and 120min during 75g oral glucose tolerance test.
  To determine whether changes in post-prandial glucagon levels correlate with changes in NEFA levels in HNF1-/4-alpha MODY patients on and off gliclazide.
Continuous glucose monitor recordings | 12 days
  To assess the blood glucose variability on and off gliclazide treatment (only for participants who opt to take part in this optional component).

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Spiliotis, MD, Principal Investigator — University of Oxford
Locations (1):
- Clinical Research Unit, OCDEM, Churchill Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The anonymised data (i.e. with studyID only) generated from this study will be deposited in the Oxford Research Archive (http://ora.ox.ac.uk/). This will provide a link between the results presented in publications and the underlying data. At the end of the retention period (currently 5 years), the data will be deleted from the archive. The anonymised data may still be used in future research.